CLINICAL TRIAL: NCT06285773
Title: The Efficacy of Recto-intercostal Fascial Plane Block and Pecto-intercostal Fascial Plane Block for Postoperative Analgesia Management After Cardiac Surgery
Brief Title: Recto-intercostal Fascial Plane Block and Pecto-intercostal Fascial Plane Block for Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 36
Record Dates: First submitted 2024-02-19; First posted 2024-02-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Disease
Keywords: Cardiac surgery; Postoperative analgesia management; Recto-intercostal fascial plane block; Pecto-intercostal fascial plane block
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification I-II and scheduled for open heart surgery (coronary artery bypass) with median sternotomy will be included in the study. Patients will be randomly divided into two groups (Group PR = PIFPB + RIFPB group, Group C = Control group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes Assessor and participant were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PR = RIFPB and PIFB group (Active Comparator): Recto-intercostal fascial plane block (RIFPB) and Pecto-intercostal fascial plane block (PIFB) will be applied
  Interventions: Drug: RIFPB block; Other: Postoperative analgesia management; Drug: PIFPB block
- Group Control (Other): No block will be applied.
  Interventions: Other: Postoperative analgesia management

INTERVENTIONS:
Drug: RIFPB block — For RIFPB, a local anesthetic will be injected into the plane between the costal cartilage and the rectus abdominis muscle at the 6th-7th costal cartilage under US guidance. The in-plane technique will be used. After confirming the block location, 10 ml of 0.25% concentration marcaine (bupivacaine) will be used (bilateral).
  Arms: Group PR = RIFPB and PIFB group
Other: Postoperative analgesia management — Patients will be administered 10mg/kg paracetamol in the postoperative period every eight hours.
  If the NRS score is ≥ 4, 1 mg kg-1 iv tramadol will be administered as a rescue analgesic.
Drug: PIFPB block — For PIFPB; the ultrasound probe for PIFB is placed 2-3 cm lateral to the upper third of the sternum, parallel to the sternum. A local anesthetic of 15 ml of 0.25% concentration of marcaine (bupivacaine) will be used between the pectoralis major and external intercostal muscles (bilateral).
  Arms: Group PR = RIFPB and PIFB group

SUMMARY:
In cardiac surgeries performed with median sternotomy, mediastinal and thoracic tube placement sites are outside the area of effect of parasternal blocks, and sometimes the sternotomy incision extends below the T6 dermatome. Recto intercostal fascial plane block (RIFPB) has been defined as a complementary block for analgesia of this region. This study aims to evaluate the effectiveness of the combination of ultrasound-guided recto-intercostal fascial plane block and pectointercostal fascial block for postoperative analgesia management after open heart surgery (coronary artery bypass) with median sternotomy.

DETAILED DESCRIPTION:
Open heart surgery is defined as surgery performed on the heart valves, arteries, and other heart structures by cutting the sternum with a median sternotomy. Cardiovascular diseases are prevalent in the general global population and affect most of the older adult population. With the increase in life expectancy in recent years, there has been a significant increase in surgical procedures for cardiovascular diseases. ERAS recommends effective perioperative pain control to improve outcomes after Cardiac Surgery. Inadequate pain control after open heart surgery causes decreased mobilization, increased respiratory complications, prolonged hospital stays, and chronic pain.

Post-heart surgery pain is most intense during the first two days and then decreases. Considering that 17% of patients report chronic pain after cardiac surgery, it is crucial to provide effective analgesia in the early postoperative period.

Failure to adequately relieve post-operative pain may lead to increased pulmonary complications as a result of inability to breathe deeply, coughing due to fear of pain, and consequent inability to clear bronchial secretions. Moreover, increased endogenous catecholamines due to surgery and pain increase the heart's oxygen consumption by causing tachycardia and hypertension. This situation causes ischemia, heart failure, and arrhythmias in patients who have undergone cardiac surgery.

In general, postoperative pain is reduced with opioids, which can cause various complications. Although the use of opioids is recommended in cardiac surgery due to their ischemic effects, multimodal perioperative pain management strategies are recommended in current anesthesia. The use of regional anesthesia as part of multimodal strategies is steadily increasing in cardiac surgeries performed through median sternotomy. Despite multimodal analgesia strategies using regional techniques, post-operative pain still emerges as an important problem in open heart surgery with median sternotomy.

The leading causes of pain after cardiac surgery are; sternotomy incisions, chest retraction, dissection of the internal mammary artery, thoracic tubes, sternal wires, and visceral pain. Sternal pain is transmitted through intercostal nerves originating from T2-T6 spinal nerve roots, whereas various regional techniques are used for analgesia in parasternal region surgeries. Amongst these techniques, while parasternal blocks can be preferred as fascial plane blocks, these aim to block the anterior cutaneous branches of the T2-T6 thoracic nerves. Pectointercostal fascial block (PIFB) is an effective technique for controlling sternal pain in heart surgeries where median sternotomy is performed.

In cardiac surgeries performed with median sternotomy, mediastinal and thoracic tube placement sites are outside the area of effect of parasternal blocks, and sometimes the sternotomy incision extends below the T6 dermatome. Recto intercostal fascial plane block (RIFPB) has been defined as a complementary block for analgesia of this region. This study aims to evaluate the effectiveness of the combination of ultrasound-guided recto-intercostal fascial plane block and pectointercostal fascial block for postoperative analgesia management after open heart surgery (coronary artery bypass) with median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-III
* Scheduled for cardiac surgery with elective median sternotomy under general anesthesia

Exclusion Criteria:

* a personal or family history of malignant hyperthermia,
* opioid sensitivity,
* alcohol or drug addiction,
* liver or kidney disease,
* skin infection in the area to be blocked,
* thoracic deformity,
* patients who are allergic to their medications,
* patients who do not agree to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Global recovery scoring system / Quality of Recovery 15 questionairre | Change from baseline score at postoperative 24 hour
  We will use the Turkish version of the Quality of Recovery / QoR-15 questionnaire. The QoR-15 ranges from 0-150 points. 0 points means the worst score, and 150 points means the best score. The QoR-15 has sections:
  Global QoR-15 Total: 150 (max) Physical Comfort 50 (max) Emotional State 40 (max) Psychological Support 20 (max) Physical Independence 20 (max) Pain 20 (max)

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Postoperative 24 hours period
  Change from Baseline Pain Scores at Postoperative 24 hours.
The use of rescue analgesia | Postoperative 24 hours period
  Tramadol using (Number of Participants using)
The use of rescue analgesia | Postoperative 24 hours period
  Tramadol using (Concentration of tramodol)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Zhang Y, Gong H, Zhan B, Chen S. Effects of bilateral Pecto-intercostal Fascial Block for perioperative pain management in patients undergoing open cardiac surgery: a prospective randomized study. BMC Anesthesiol. 2021 Jun 22;21(1):175. doi: 10.1186/s12871-021-01391-w. PMID 34157970
- [Background] Khera T, Murugappan KR, Leibowitz A, Bareli N, Shankar P, Gilleland S, Wilson K, Oren-Grinberg A, Novack V, Venkatachalam S, Rangasamy V, Subramaniam B. Ultrasound-Guided Pecto-Intercostal Fascial Block for Postoperative Pain Management in Cardiac Surgery: A Prospective, Randomized, Placebo-Controlled Trial. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):896-903. doi: 10.1053/j.jvca.2020.07.058. Epub 2020 Jul 24. PMID 32798172
- [Background] Elbardan IM, Shehab AS, Mabrouk IM. Comparison of Transversus Thoracis Muscle Plane Block and Pecto-Intercostal Fascial Plane Block for enhanced recovery after pediatric open-heart surgery. Anaesth Crit Care Pain Med. 2023 Aug;42(4):101230. doi: 10.1016/j.accpm.2023.101230. Epub 2023 Apr 7. PMID 37031816
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Alver S, Sakul BU, Ansen G, Pence KB, Alici HA. Recto-intercostal fascial plane block: Another novel fascial plane block. J Clin Anesth. 2023 Oct;89:111163. doi: 10.1016/j.jclinane.2023.111163. Epub 2023 Jun 7. No abstract available. PMID 37295124